CLINICAL TRIAL: NCT06959342
Title: Modification of Inhibitory Control and Craving Through Transcranial Direct Current Stimulation (tDCS) as an Add-On Treatment for Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Wellcome Leap Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-561N-MA
Record Dates: First submitted 2025-04-02; First posted 2025-05-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder; Substance Use Disorders
Keywords: Transcranial Direct Current Stimulation; tDCS; Inhibition Training; Electroencephalography; EEG; Inhibitory Control; Working Memory; Craving
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding of the tDCS stimulation groups: Participants do not receive any information about electrode placement or active vs. sham condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- right dlPFC (Experimental): tDCS anodal electrode over the right dlPFC (position F4, EEG cap 10/20 system), cathodal electrode over the left dlPFC (position F3, EEG cap 10/20 system).
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- left dlPFC (Active Comparator): tDCS anodal electrode over the left dlPFC (position F3, EEG cap 10/20 system), cathodal electrode over the right dlPFC (position F4, EEG cap 10/20 system).
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Occipital Cortex (Active Comparator): tDCS anodal electrode over the occipital cortex (position O1, EEG cap 10/20 system), cathodal electrode over position Cz (EEG cap 10/20 system).
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): tDCS anodal electrode over the right dlPFC (position F4, EEG cap 10/20 system), cathodal electrode over the left dlPFC (position F3, EEG cap 10/20 system). The current is ramped up from 0.3mA to initially 2mA (0.1mA/s) and then immediately ramped down.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Computerized Inhibition Training (Active Comparator): Standardized computerized inhibition training using a go-/no-go-task with individually adapted, substance-related stimuli (wine, beer, spirits).
  Interventions: Behavioral: Inhibition Training
- Treatment as Usual (No Intervention): Patients only receive standard treatment in clinic (qualified detoxification program).

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — tDCS sessions on five consecutive days for 20 minutes.
  Other Names: Sooma Medical
  Arms: Occipital Cortex; Sham tDCS; left dlPFC; right dlPFC
Behavioral: Inhibition Training — Computerized Training of inhibitory control (Go-/No-Go task with pictures of preferred alcohol) on five consecutive days.
  Arms: Computerized Inhibition Training

SUMMARY:
The aim of this project is to investigate the potential of transcranial direct current stimulation (tDCS) to reduce cognitive deficits and substance craving in individuals with substance use disorders (SUD), with a focus on alcohol use disorder (AUD). Patients of any gender between the ages of 18 and 65 are examined who are in our inpatient and day clinic settings for a standard detoxification treatment program. As there are conflicting findings regarding the effective settings for tDCS as an adjunctive treatment in SUD (e.g., effects on inhibitory control seem to be sensitive to current direction), the aim is to examine and compare three different active tDCS conditions, a sham tDCS condition (placebo), inhibition training, and a control group of patients receiving only standard detoxification treatment. The aim is to identify the optimal electrode placement and current direction to positively influence both inhibitory control and craving, leading to improved treatment outcomes such as longer abstinence periods or reduced substance use after relapse.

DETAILED DESCRIPTION:
The aim of this study is to determine the optimal electrode placement and current direction of tDCS as an adjunctive therapy for SUD to improve both inhibitory control and craving, ultimately contributing to better treatment outcomes such as longer abstinence periods and reduced substance use after relapse. To achieve this, the investigators will assess inhibitory control in SUD patients using computerized neuropsychological testing before and after multiple tDCS sessions with different stimulation protocols. In addition, the effects of tDCS on inhibitory control will be investigated by EEG recordings, focusing on the N2 and P3 components.

To ensure that tDCS stimulation occurs at exactly the same location for each stimulation session, tDCS electrodes (25 cm2) are placed at defined locations in the EEG cap (10/20 system) using saline-soaked sponges. The current is ramped up from 0.3 mA to 2 mA at a rate of 0.1 mA per second and remains at 2 mA for the duration of the active stimulation (20 min total; 0.08 mA/cm2). The tDCS sessions last 20 minutes on five consecutive days.

Four active tDCS stimulations, one sham stimulation, two active control groups and one control group without ad-on treatment are investigated. All groups receive a qualified detoxification treatment in the clinic. First, the investigators want to test whether anodal stimulation is indeed hemispherically sensitive in affecting inhibitory control, while craving reduction is independent of it. Since tDCS (with one anodal and one cathodal electrode) has a poor spatial resolution, the investigators also want to test whether tDCS has a more general effect on brain metabolism and thus on task performance. Therefore, the study includes a control group with anodal stimulation over the occipital cortex at the border with the cerebellum. In addition, computerized inhibition training will be performed to investigate the effects of active, high-frequency contact and behavioral training compared to tDCS. Participants will also receive the same protocol with sham tDCS as well as a no-intervention group to avoid confounding by placebo effects and to control whether participation in the study itself constitutes a "treatment".

On the first examination day (T1), psychometric measures are collected, neuropsychological testing is conducted, and EEG recordings are performed during a modified Go/No-Go task. Depending on group allocation, participants receive their first tDCS session, inhibition training, sham stimulation, or no intervention. On intervention days 2-4 (T2-T4), participants continue their assigned interventions. On day 5 (T5), they receive the final intervention along with another EEG measurement during the Go/No-Go task. Follow-up assessments take place via telephone at 4 weeks (T6), 8 weeks (T7), and 24 weeks (T9) to record self-reported relapse and substance use. At 12 weeks (T8), participants return for an in-person assessment, including EEG measurement during the modified Go/No-Go task.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis: alcohol use disorder according to DSM-5
* patients of any gender aged 18 to 65
* normal vision or correctable visual impairment.
* sufficient ability to communicate verbally and in writing
* ability to give fully informed consent after reviewing thorough written information

Exclusion Criteria:

* withdrawal of consent
* severe internal, neurological, or psychiatric comorbidities (e.g., lifetime schizophrenia, bipolar disorder, or other severe mental disorders according to ICD-10 and DSM-5, such as severe depression or PTSD within the last 12 months).
* Exclusion criteria for an EEG/tDCS examination (e.g. metal implants in the head, epilepsy, etc.)
* severe withdrawal symptoms (CIWA-R > 7)
* alcohol intoxication (breath alcohol concentration > 0 ‰)
* Pharmacotherapy with psychoactive substances within the last 14 days (exceptions: clomethiazole or benzodiazepines used in withdrawal treatment, provided they were discontinued at least 3 days prior; antidepressants or anxiolytics taken at stable doses).
* drug or alcohol use within the last 7 days
* for women: pregnancy
* suicidal tendencies or danger to others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Inhibitory Control (Go/No-Go Task) | intervention day 1 (T1), intervention day 5 (T5), follow-up after 12 weeks (T8)
  Change in performance in a modified Go/No-Go task. Measures inhibitory control under varying working memory loads.
Inhibitory Control (EEG) | intervention day 1 (T1), intervention day 5 (T5), follow-up after 12 weeks (T8)
  Change in event-related potentials (ERPs), specifically the P300 and N200 components, measured by EEG during Go-/NO-GO task (32 channels with active electrodes, mBrainTrain, Belgrade, Serbia); sampling rate 1000Hz, filtered between 0.016-1000Hz, programmed in Presentation® software (Neurobehavioral Systems, Inc., Berkeley, CA, USA).
Craving | intervention day 1 and 5 (T1, T5), follow-up after 4 weeks (T6), follow-up after 8 weeks (T7), follow-up after 12 weeks (T8), follow-up after 24 weeks (T9)
  Change in subjective craving according to Alcohol Urge Questionnaire and craving scale.
  Alcohol Urge Questionnaire: 7-item Likert scale ranging from "strongly disagree" to "strongly agree"). A total score is calculated by averaging the scores for each item. Higher scores indicate stronger craving.
  Craving scale: Craving from 0-100%. Higher scores indicate stronger cravings.

SECONDARY OUTCOMES:
Relapse/Alcohol Use | intervention day 1 and 5 (T1, T5), follow-up after 4 weeks (T6), follow-up after 8 weeks (T7), follow-up after 12 weeks (T8), follow-up after 24 weeks (T9)
  Change in number of drinking days, number of abstinent days, number of days with more than 48/60g (women/men) of alcohol, cumulative amount of alcohol in grams.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Central Institute of Mental Health, Mannheim
  - Psychiatrisches Zentrum Nordbaden (Psychiatric Center Nordbaden), Wiesloch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stock AK, Riegler L, Chmielewski WX, Beste C. Paradox effects of binge drinking on response inhibition processes depending on mental workload. Arch Toxicol. 2016 Jun;90(6):1429-36. doi: 10.1007/s00204-015-1565-y. Epub 2015 Jul 1. PMID 26126633
- [Background] Stein M, Soravia LM, Tschuemperlin RM, Batschelet HM, Jaeger J, Roesner S, Keller A, Gomez Penedo JM, Wiers RW, Moggi F. Alcohol-specific inhibition training in patients with alcohol use disorder: a multi-centre, double-blind randomized clinical trial examining drinking outcome and working mechanisms. Addiction. 2023 Apr;118(4):646-657. doi: 10.1111/add.16104. Epub 2023 Jan 3. PMID 36468408
- [Derived] Vollstadt-Klein S, Turkmen C, Grundinger N, Wieland A, Aggensteiner PM, Stock AK, Stein M, Moggi F, Bublatzky F, Kiefer F, Link T, Gerhardt S. Modification of inhibitory control and craving through transcranial direct current stimulation as an add-on treatment for substance use disorder: protocol for a randomized controlled study. BMC Psychol. 2025 Oct 13;13(1):1132. doi: 10.1186/s40359-025-03506-1. PMID 41084082